CLINICAL TRIAL: NCT07099963
Title: Frequency and Severity of Respiratory Acidosis During One-lung Ventilation, a Retrospective Pilot Study to Compare Clinician Settings and Those Proposed by the VentilO Application
Status: Recruiting | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, François Lellouche, Principal Investigator, Laval University
Other Study IDs: 2026-4405
Record Dates: First submitted 2025-07-02; First posted 2025-08-01 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Thoracic; Surgery; Mechanical Ventilation; Hypercapnia; Acidosis; One Lung Ventillation (OLV); Smartphone Application
MeSH Terms: conditions — Hypercapnia; Acidosis | interventions — One-Lung Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Thoracic surgery: Patient managed with one lung ventilation
  Interventions: Other: one lung ventilation

INTERVENTIONS:
Other: one lung ventilation — Arterial blood gases during one lung ventilation

SUMMARY:
One-lung ventilation is a mechanical ventilation method frequently used during several thoracic surgeries. One-lung ventilation requires the use of protective ventilation to limit ventilator-induced injury and reduce postoperative respiratory complications. Protective ventilation during one-lung ventilation is specific since tidal volumes are applied by definition to one lung, and it is recommended to use lower tidal volumes, down to 4 ml/kg of ideal body weight. This approach requires individualized ventilation parameters, which differs from the conventional or two-lung ventilation, and there are no clear recommendations regarding respiratory rate adjustment to ensure adequate gas exchange.

DETAILED DESCRIPTION:
The aim of the study is to:

1. Evaluate whether the initial ventilation settings (tidal volume and respiratory rate) during one-lung ventilation are appropriate to prevent respiratory acidosis.
2. Compare the ventilation settings (tidal volume and respiratory rate) made by clinicians with those proposed by an smartphone application ''VentilO''.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years old)
* Patients intubated and undergoing one-lung ventilation during thoracic surgery
* Volume-controlled ventilation mode used intraoperatively

Exclusion Criteria:

* Arterial blood gas data unavailable during one-lung ventilation
* Missing demographic data (sex, height, actual weight)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient undergoing thoracic surgery requiring intraoperative one-lung ventilation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Respiratory acidosis | 20 minutes after initiation of one lung ventilation after lung isolation
  The frequency of respiratory acidosis on arterial blood gases after 20 minutes of mechanical ventilation (pH < 7.35 and PaCO2 > 45mmHg) measured by arterial blood gases

SECONDARY OUTCOMES:
Respiratory rate | At the beginning of one lung ventilation during the surgery
  Respiratory rate set by the doctor, this respiratory rate will be compared to the suggestion of the algorithm
Acid-base disorder | At the beginning of one lung ventilation during the surgery
  Presence of Respiratory alkalosis define by pH>7.45 and PaCO2 < 35 mmHg
Number of participants with hemodynamic shock - hypotension | Day 1
  Requiring >1L of volume repletion and/or use of amines at >0.05 mcg/kg/min or norepinephrine equivalent
Hospital length of stay | Up to 90 days
  Recovery room admission through hospital discharge
Mechanical Ventilation duration | Up to 90 days
  Time spent with invasive mechanical ventilation during surgery and hospital stay
Hospital mortality | Up to 90 days
  Occurence of death during hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec - Université Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No